CLINICAL TRIAL: NCT04026165
Title: MOSAIC - A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study Evaluating the Efficacy and Safety of Selonsertib in Subjects With Moderate to Advanced Diabetic Kidney Disease
Brief Title: Study to Evaluate the Efficacy and Safety of Selonsertib in Participants With Moderate to Advanced Diabetic Kidney Disease
Acronym: MOSAIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-223-1017; JapicCTI-194911 (Registry Identifier: Japan Pharmaceutical Information Center); 2018-003951-39 (EudraCT Number)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: Participants received Run-in and Randomized treatments sequentially and in the Randomized Phase, the treatments were assigned in parallel.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selonsertib (Experimental): Run-in Period (5 Weeks): Participants will receive placebo-to-match SEL for at least one week and then SEL 18 mg for at least 4 weeks.
  Randomized Period: Participants will be randomized to receive SEL 18 mg for at least 48 weeks.
  Interventions: Drug: SEL; Drug: Placebo
- Placebo (Placebo Comparator): Run-in Period (5 Weeks): Participants will receive placebo-to-match SEL for at least one week and then SEL 18 mg for at least 4 weeks.
  Randomized Period: Participants will be randomized to receive placebo-to-match SEL for at least 48 weeks.
  Interventions: Drug: SEL; Drug: Placebo

INTERVENTIONS:
Drug: SEL — Tablet administered orally once daily
Drug: Placebo — Tablet administered orally once daily

SUMMARY:
The primary objective of this study is to evaluate whether selonsertib (SEL) can slow the decline in kidney function in participants with moderate to advanced diabetic kidney disease (DKD).

DETAILED DESCRIPTION:
Following the screening period, eligible participants will enroll into a Run-in period of at least 5 weeks and receive placebo to match SEL for at least 1 week and then SEL for at least 4 weeks. After completing Run-in period, eligible participants will be randomized and receive either SEL or placebo to match SEL for at least 48 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (T2DM) as per local guidelines.
* Estimated glomerular filtration rate (eGFR) value calculated by central laboratory utilizing samples collected during screening and prior to enrollment of ≥ 20 mL/min/1.73 m^2 to < 60 mL/min/1.73 m^2 with albuminuria

  * eGFR and urine albumin to creatinine ratio (UACR) must meet criteria a, b, or c

    * a: eGFR (mL/min/1.73 m^2): ≥ 45 to < 60; UACR (mg/g): ≥ 600 to 5000
    * b: eGFR (mL/min/1.73 m^2): ≥ 30 to < 45; UACR (mg/g): ≥ 300 to 5000
    * c: eGFR (mL/min/1.73 m^2): ≥ 20 to < 30; UACR (mg/g): ≥ 150 to 5000
* Treatment with either an angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB)

  * Individuals not receiving an ACEi or ARB may be enrolled if there is documented intolerance to ACEi and ARB
  * Individuals receiving less-than-maximal dose of an ACEi or ARB may be enrolled if there is a documented reason that the maximum labeled dose of ACEi and ARB could not be reached
* Individuals already receiving sodium-glucose co-transporter-2 (SGLT-2) inhibitors must be on a stable dose for at least 2 weeks prior to enrollment
* Mean systolic blood pressure (SBP) must be <160 mmHg and mean diastolic blood pressure (DBP) must be <100 mmHg
* Required baseline laboratory data, analyzed by central laboratory, within 30 days prior to enrollment

Key Exclusion Criteria:

* Hemoglobin A1c (HbA1c) > 12.0% within 30 days prior to enrollment
* Individuals with diagnosis of type 1 diabetes mellitus (T1DM) or maturity onset diabetes of the young (MODY)
* Body mass index (BMI) > 50 kg/m^2
* UACR > 5000 mg/g on any measurement during screening
* End stage kidney disease (ESKD) (i.e., chronic hemodialysis, chronic peritoneal dialysis, or history of kidney transplantation)
* Anticipated progression to ESKD (need for chronic hemodialysis, chronic peritoneal dialysis or receipt of kidney transplant) within 3 months after enrollment
* Unstable cardiovascular disease
* Pregnant or lactating females or planning to become pregnant or breastfeed during the study
* Concurrent use of either

  1. ACEi and ARB or
  2. Mineralocorticoid receptor antagonist (MRA) or direct renin inhibitor (DRI) in combination with an ACEi or ARB for at least 2 weeks prior to Enrollment
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the individual or impair the assessment of study results

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (111):
- United States (71):
  - Arizona Kidney Disease and Hypertension Centers, Glendale, Arizona
  - AKDHC Medical Research Services, LLC, Tucson, Arizona
  - Clearview Medical Research, LLC, Canyon Country, California
  - Kidney Disease Medical Group, Inc., Glendale, California
  - Renal Consultants Medical Group, Granada Hills, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - California Institute of Renal Research, La Mesa, California
  - Academic Medical Research Institute, Los Angeles, California
  - Rose Salter Medical Research Foundation, Newport Beach, California
  - Valley Renal Medical Group Research, Northridge, California
  - California Institute of Renal Research, San Diego, California
  - California Kidney Specialist, San Dimas, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - New West Physicians, Inc, Golden, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC, Westminster, Colorado
  - Omega Research Maitland, LLC, DeBary, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Discovery Medical Research Group, Inc, Ocala, Florida
  - Coastal Nephrology Associates Research Center, LLC. D/B/A Volunteer Medical Research, Port Charlotte, Florida
  - Atlanta Center for Clinical Research, Atlanta, Georgia
  - Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Boise Kidney & Hypertension, PLLC, Meridian, Idaho
  - Research By Design, LLC, Chicago, Illinois
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Internal Medicine Specialists, Inc, New Orleans, Louisiana
  - Northwest Louisiana Nephrology L.L.C, Shreveport, Louisiana
  - Aa Mrc, Llc, Flint, Michigan
  - Elite Research Center, Flint, Michigan
  - Arcturus Healthcare, PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Pelican Point Dialysis - DaVita Clinical Research, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - North Shore University Hospital: Division of Nephrology, Great Neck, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - CHEAR Center LLC, The Bronx, New York
  - Mountain Kidney and Hypertension Associates, Asheville, North Carolina
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Diabetes And Endocrinology Consultants, P.C., Morehead City, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research Inc., d/b/a PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - SV Research LLC, Marion, Ohio
  - Midwest Nephrology Group, PLLC, Midwest City, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Lifespan Clinical Research Center, East Providence, Rhode Island
  - PMG Research Of Charleston, LLC, Mt. Pleasant, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - PMG Research, Inc d/b/a/ PMG Research of Knoxville, Knoxville, Tennessee
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - PMG Research, Inc. d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Memphis Veteran Affairs Medical Center, Memphis, Tennessee
  - Arlington Nephrology, Arlington, Texas
  - Corsicana Medical Research, LLC, Corsicana, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - The Medical Group of Texas, Fort Worth, Texas
  - Primecare Medical Group, Houston, Texas
  - DaVita Clinical Research, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - DaVita Clinical Research, Lewisville, Texas
  - Houston Methodist Research Institute - CCAT Pearland, Pearland, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
- Australia (3):
  - Austin Health and University of Melbourne, Heidelberg, Victoria
  - St. Vincent Hospital, Melbourne, Fitzroy
  - Royal Melbourne Hospital, Parkville
- Canada (8):
  - LMC Clinical Research Inc. (Barrie), Barrie
  - LMC Clinical Research Inc. (Brampton), Brampton
  - LMC Clinical research Inc. (Thornhill), Concord
  - LMC Clinical Research Inc. (Etobicoke), Etobicoke
  - Clinical Research Solution Inc., Kitchener
  - Centre de Recherche Clinique de Lava, Laval
  - Dr TGElliott Inc dba BC Diabetes, Vancouver
  - Winnipeg Clinic, Winnipeg
- Japan (24):
  - Asahikawa Medical University Hospital, Asahikawa
  - National Hospital Organization Chiba-East-Hospital, Chiba
  - Kagoshima University Hospital, Kagoshima
  - Kokura Memorial Hospital, Kitakyushu-shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurobe City Hospital, Kurobe-shi
  - Kurume University Hospital, Kurume-shi
  - Nakamoto Medical Clinic, Mito
  - Kozawa Eye Hospital and Diabetes Center, Mito
  - Japanese Red Cross Musashino Hospital, Musashino
  - Nagasaki University Hospital, Nagasaki
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital, Nagoya
  - Daido Clinic, Nagoya
  - Nakakinen Clinic, Naka
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka General Medical Center, Osaka
  - Hoshina Clinic, Saitama-shi
  - Sanuki Municipal Hospital, Sanuki-shi
  - Tachikawa Hospital, Tachikawa-shi
  - Mishuku Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - TOYOTA Memorial Hospital, Toyota-shi
  - Yokohama City University Hospital, Yokohama
- New Zealand (5):
  - Auckland City Hospital (Auckland District Health Board), Auckland
  - Middlemore Clinical Trials Trust trading as Middlemore Clinical Trials, Auckland
  - Lipid and Diabetes Research Group, Christchurch
  - Waitemata District Health Board- North Shore Hospital, North Shore
  - Endocrine, Diabetes & Research Centre (Capital and Coast District Health Board), Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heerspink HJL, Perkovic V, Tuttle KR, Pergola PE, Mahaffey KW, Patel UD, Ishida JH, Kuo A, Chen F, Kustra R, Petrovic V, Rossing P, Kashihara N, Chertow GM. Selonsertib in Patients with Diabetic Kidney Disease: A Phase 2b Randomized Active Run-In Clinical Trial. J Am Soc Nephrol. 2024 Dec 1;35(12):1726-1736. doi: 10.1681/ASN.0000000000000444. Epub 2024 Jul 17. PMID 39018154
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-223-1017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Japan, Canada, New Zealand, and Australia.
Pre-assignment Details: 961 participants were screened.
Groups:
- Run-in Placebo: Participants received placebo to match selonsertib (SEL) tablet orally once daily for at least one week.
- Run-in SEL 18 mg: Participants received SEL 18 mg tablet orally once daily for at least 4 weeks.
- Randomized SEL 18 mg: Participants received SEL 18 mg tablet orally once daily for at least 4 weeks in the Run-in period, were then randomized, and received SEL 18 mg tablet orally once daily for at least 48 weeks.
- Randomized Placebo: Participants received SEL 18 mg tablet orally once daily for at least 4 weeks in the Run-in period, were then randomized, and received placebo-to-match SEL tablet orally once daily for at least 48 weeks.
Period: Run-in Placebo Period
Arm/Group | Run-in Placebo | Run-in SEL 18 mg | Randomized SEL 18 mg | Randomized Placebo
Started | 384 (Following the screening period, eligible participants were enrolled into Run-in Placebo period for at least one week.) | 0 | 0 | 0
Completed | 362 | 0 | 0 | 0
Not Completed | 22 | 0 | 0 | 0
Not completed — Enrollment Error | 13 | 0 | 0 | 0
Not completed — Run-in Failure | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Withdrew Consent | 2 | 0 | 0 | 0
Not completed — Significant Non-Compliance with Study Drug | 1 | 0 | 0 | 0
Period: Run-in SEL Period
Arm/Group | Run-in Placebo | Run-in SEL 18 mg | Randomized SEL 18 mg | Randomized Placebo
Started | 0 (Following the Run-in Placebo period, participants took SEL (18 mg) for at least 4 weeks in Run-in SEL period.) | 357 (Following the Run-in Placebo period, participants took SEL (18 mg) for at least 4 weeks in Run-in SEL period.) | 0 | 0
Completed | 0 | 311 | 0 | 0
Not Completed | 0 | 46 | 0 | 0
Not completed — Run-in Failure | 0 | 26 | 0 | 0
Not completed — Withdrew Consent | 0 | 10 | 0 | 0
Not completed — Enrollment Error | 0 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0
Not completed — Investigator's Discretion | 0 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: Randomized Period
Arm/Group | Run-in Placebo | Run-in SEL 18 mg | Randomized SEL 18 mg | Randomized Placebo
Started | 0 | 0 (Following the Run-in period, eligible participants were randomized to receive either SEL (18 mg) or placebo.) | 154 (Following the Run-in period, eligible participants were randomized to receive either SEL (18 mg) or placebo.) | 156 (Following the Run-in period, eligible participants were randomized to receive either SEL (18 mg) or placebo.)
Completed | 0 | 0 | 140 | 137
Not Completed | 0 | 0 | 14 | 19
Not completed — Withdrew Consent | 0 | 0 | 5 | 8
Not completed — Death | 0 | 0 | 5 | 7
Not completed — Investigator's Discretion | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of Run-in SEL.
Groups:
- Run-in SEL 18 mg, Not Randomized: Participants received SEL 18 mg tablet orally once daily for at least 4 weeks in the Run-in period and were not randomized.
- Total: Total of all reporting groups
Arm/Group | Run-in SEL 18 mg, Not Randomized | Randomized SEL 18 mg | Randomized Placebo | Total
Number analyzed (Participants) | 47 | 154 | 156 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.7) | 65 (9.3) | 66 (8.8) | 65 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 48 | 51 | 111
  Male | 35 | 106 | 105 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 132 | 136 | 307
  Not Hispanic or Latino | 8 | 21 | 19 | 48
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 2 | 0 | 2
  Race: Asian | 4 | 41 | 44 | 89
  Race: Black or African American | 4 | 26 | 22 | 52
  Race: Native Hawaiian or Pacific Islander | 1 | 5 | 4 | 10
  Race: White | 36 | 78 | 84 | 198
  Race: Other | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  New Zealand | 0 | 7 | 8 | 15
  Canada | 8 | 11 | 9 | 28
  United States | 38 | 96 | 99 | 233
  Japan | 1 | 38 | 37 | 76
  Australia | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Treatment-specific Baseline Estimated Glomerular Filtration Rate Based on Creatinine (eGFRcr)
Description: The values of eGFRcr were calculated using the Chronic Kidney Disease Epidemiology (CKD-EPI) Creatinine Equation (2009). eGFRcr = 141*min(Standardized Serum Creatinine (Scr)/kappa, 1) ^alpha*max(Scr/ kappa, 1)^(-1.209)*0.993^Age*1.018[if female]*1.159[if Black], where kappa=0.7(females) or 0.9(males), alpha=-0.329(females) or -0.411(males). min indicates the minimum of Scr/kappa or 1, max indicates the maximum of Scr/kappa or 1, and age is in years.
  Treatment-specific Baselines = the average of Visits A and B values for Placebo, and the average of Visit C and Day 1 values for SEL.
  Visit A= enrollment, Visit B= 7-14 days after Visit A, Visit C= 21-28 days after Visit B, and Visit 1= 7-14 days after Visit C.
Time Frame: Treatment-specific Baselines (From enrollment (Visit A) up to 14 days after Visit A for placebo and from Visit C up to 14 days after Visit C for SEL)
Population: The Full Analysis Set included all participants who were randomized in the study, and received at least one dose of study drug in the Randomization Phase.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Randomized SEL 18 mg | Randomized Placebo
Number analyzed (Participants) | 154 | 156
mL/min/1.73m^2 | 32.7 (10.59) | 34.9 (10.81)

2. Primary Outcome: eGFRcr Slope
Description: The values of eGFRcr were calculated using the CKD-EPI Creatinine Equation (2009). eGFRcr = 141*min(Scr/kappa, 1) ^alpha*max(Scr/kappa, 1)^(-1.209)*0.993^Age*1.018[if female]*1.159[if Black], where kappa=0.7(females) or 0.9(males), alpha=-0.329(females) or -0.411(males). min indicates the minimum of Scr/kappa or 1, max indicates the maximum of Scr/kappa or 1, and age is in years. Treatment specific baselines for eGFRcr: average of Visit A (enrollment) and Visit B (7-14 days after Visit A) values for Placebo, and average of Visit C (21-28 days after Visit B, and Visit 1 (7-14 days after Visit C) values for SEL.
Time Frame: Treatment-specific Baselines through Week 84
Population: Participants in the Full Analysis Set (included all participants who were randomized in the study and received at least 1 dose of study drug in the randomization phase) with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2/year
Arm/Group | Randomized SEL 18 mg | Randomized Placebo
Number analyzed (Participants) | 153 | 156
mL/min/1.73m^2/year | -2.29 (0.58) | -3.49 (0.58)
Statistical Analysis 1: Comparison: Randomized SEL 18 mg vs Randomized Placebo; Estimates were from a random slope model with change in eGFRcr from treatment-specific Baselines at Weeks 4, 8, 12, 24, 36, 48, 60, 72, and 84 as outcome, including terms for treatment-specific Baseline eGFRcr, pre-run-in urine albumin to creatinine ratio (UACR) category (< 1500 mg/g vs. >= 1500 mg/g), concomitant use of sodium-glucose co-transporter-2 (SGLT-2) inhibitors at Randomization, treatment group, week, and treatment-by-week interaction, where week has a random effect; Test type: Superiority; p = 0.1439, Random Slope Model; Difference in Adjusted Mean = 1.20, 95% CI 2-sided [-0.41 to 2.81], Standard Error of Mean 0.82

3. Secondary Outcome: Percentage of Participants With Kidney Clinical Events at Week 48
Description: Kidney clinical events were defined as any of the following events: confirmed ≥ 40% decline in eGFRcr from baseline, or kidney failure (dialysis performed for at least 4 weeks, kidney transplantation, or confirmed decrease in eGFRcr to < 15 mL/min/1.73 m^2 for participants without dialysis or kidney transplantation), or death due to kidney disease.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized SEL 18 mg | Randomized Placebo
Number analyzed (Participants) | 154 | 156
percentage of participants | 9.1 | 9.0
Statistical Analysis 1: Comparison: Randomized SEL 18 mg vs Randomized Placebo; Test type: Superiority; p = 0.8353, Cochran-Mantel-Haenszel — p-value was based on Cochran-Mantel-Haenszel test stratified by Randomization stratification factors. Randomization stratification factors= pre-run-in eGFRcr stratum, pre-run-in UACR category and concomitant use of SGLT-2 inhibitors at Randomization; Difference in Percentage = 0.1, 95% CI 2-sided [-10.9 to 11.4] — 95% exact CI based on the Santner-Snell method was presented for the difference in proportions between SEL and placebo arms

4. Secondary Outcome: Time From Randomization to First Occurrence of a Kidney Clinical Event: Event Rate Per 100 Participant-years for First Occurrence of Kidney Clinical Event
Description: Kidney clinical events were defined as any of the following events: confirmed ≥ 40% decline in eGFRcr from baseline, or kidney failure (dialysis performed for at least 4 weeks, kidney transplantation, or confirmed decrease in eGFRcr to < 15 mL/min/1.73 m^2 for participants without dialysis or kidney transplantation), or death due to kidney disease. This outcome measure was analyzed using event rate per 100 participant-years for first occurrence of kidney clinical event. Participant year was calculated as total follow-up duration across all participants in a given group. Follow-up duration was defined as time from Randomization to the earliest of study completion, premature study discontinuation, death, or event of interest in each row.
Time Frame: From randomization up to Week 101
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: events per 100 participant-years
Arm/Group | Randomized SEL 18 mg | Randomized Placebo
Number analyzed (Participants) | 154 | 156
events per 100 participant-years | 13.4 | 9.8
Statistical Analysis 1: Comparison: Randomized SEL 18 mg vs Randomized Placebo; Test type: Superiority; p = 0.2010, Stratified Log-Rank; P-value was calculated using a stratified log-rank test, stratified by randomization stratification factors; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [0.81 to 2.72] — Hazard ratio and 95% CI were estimated using a stratified Cox proportional hazard model, stratified by randomization stratification factors and were reported only for outcomes with more than 10 events, and have at least 1 event in each treatment arm

5. Secondary Outcome: Pre-run-in Baseline Estimated Glomerular Filtration Rate Based on Cystatin C (eGFRcys)
Description: eGFRcys = Estimated Glomerular Filtration Rate calculated by CKD-EPI Cystatin C Equation (2012). eGFR = 133*min(Standardized Serum Cystatin (Scys)/0.8, 1) ^(-0.499)*max(Scys/0.8, 1)^(-1.328)*0.996^Age*0.932[if female]. min indicates the minimum of Scys/0.8 or 1, max indicates the maximum of Scr/0.8 or 1, and age is in years.
Time Frame: Pre-run-in Baseline (Pre-run in Baseline = Average of visit A (Enrollment) and Visit B (7-14 days after Visit A) eGFRcys values)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Randomized SEL 18 mg | Randomized Placebo
Number analyzed (Participants) | 154 | 156
mL/min/1.73m^2 | 33.6 (11.81) | 32.4 (10.94)

6. Secondary Outcome: eGFRcys Slope
Description: eGFRcys = Estimated Glomerular Filtration Rate calculated by CKD-EPI Cystatin C Equation (2012). eGFR = 133*min(Scys/0.8, 1) ^(-0.499)*max(Scys/0.8, 1)^(-1.328)*0.996^Age*0.932[if female]. min indicates the minimum of Scys/0.8 or 1, max indicates the maximum of Scr/0.8 or 1, and age is in years. Pre-run in Baseline = Average of visit A (Enrollment) and Visit B (7-14 days after Visit A) eGFRcys values.
Time Frame: Pre-run-in Baseline through Week 84
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2/year
Arm/Group | Randomized SEL 18 mg | Randomized Placebo
Number analyzed (Participants) | 153 | 156
mL/min/1.73m^2/year | -3.79 (0.51) | -4.23 (0.51)
Statistical Analysis 1: Comparison: Randomized SEL 18 mg vs Randomized Placebo; Estimates were from a random slope model with change in eGFRcys from pre-run-in Baseline at Weeks 4, 8, 12, 24, 36, 48, 60, 72, and 84 as outcome, including terms for pre-run-in Baseline eGFRcys, pre-run-in UACR category (< 1500 mg/g vs. >= 1500 mg/g), concomitant use of SGLT-2 inhibitors at Randomization, treatment group, week, and treatment-by-week interaction, where week has a random effect; Test type: Superiority; p = 0.5399, Random Slope Model; Difference in Adjusted Mean = 0.44, 95% CI 2-sided [-0.97 to 1.86], Standard Error of Mean 0.72

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to maximum duration of 107.1 weeks; Adverse Events: First dose in Run-in SEL phase up to last dose (maximum: 101 weeks) plus 30 days
Description: All-Cause Mortality: The All Enrolled Analysis Set included all participants who were enrolled in the study.
  Adverse Events: The Safety Analysis Set included all participants who took at least 1 dose of Run-in SEL.
Groups:
- Run-in Placebo: Participants received placebo-to-match SEL tablet orally once daily for at least one week.
- Randomized SEL 18 mg: Participants received SEL 18 mg tablet orally once daily for at least 48 weeks after Randomization.
- Randomized Placebo: Participants received placebo-to-match SEL tablet orally once daily for at least 48 weeks after Randomization.
Arm/Group | Run-in Placebo | Run-in SEL 18 mg | Randomized SEL 18 mg | Randomized Placebo
All-Cause Mortality (participants affected / at risk) | 0/384 | 1/357 | 5/154 | 7/156
Serious Adverse Events (participants affected / at risk) | 0/0 | 16/357 | 45/154 | 45/156
Other Adverse Events (participants affected / at risk) | 0/0 | 37/357 | 55/154 | 49/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Placebo (N=0) | Run-in SEL 18 mg (N=357) | Randomized SEL 18 mg (N=154) | Randomized Placebo (N=156)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 5
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 3 | 3 | 5
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 2
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 5 | 2
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 5 | 3
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arteriogram coronary abnormal (Investigations) | 0 | 0 | 1 | 0
Carbon dioxide abnormal (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Device end of service (Product Issues) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 10 | 7
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 3
Renal mass (Renal and urinary disorders) | 0 | 0 | 1 | 0
Subcapsular renal haematoma (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Placebo (N=0) | Run-in SEL 18 mg (N=357) | Randomized SEL 18 mg (N=154) | Randomized Placebo (N=156)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 5 | 8
Constipation (Gastrointestinal disorders) | 0 | 7 | 11 | 3
Oedema peripheral (General disorders) | 0 | 5 | 11 | 8
Urinary tract infection (Infections and infestations) | 0 | 6 | 5 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 8 | 12 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 6 | 9
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 10 | 4
Hypertension (Vascular disorders) | 0 | 10 | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT04026165/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT04026165/SAP_001.pdf